CLINICAL TRIAL: NCT01449292
Title: Study of the AeriSeal System for HyPerInflation Reduction in Emphysema (ASPIRE)
Acronym: ASPIRE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-C11-003PLV
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Pulmonary Emphysema
Keywords: PLVR; ELVR; AeriSeal System; foam sealant; emphysematous lung sealant; ELS; COPD; emphysema; polymeric lung volume reduction; heterogeneous; Respiratory Tract Diseases; Lung Diseases; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Emphysema; Pulmonary Disease, Chronic Obstructive; Emphysema; Respiratory Tract Diseases; Lung Diseases | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment plus Optimal Medical Therapy (Experimental): Patients will be treated with the AeriSeal System and Optimal Medical Therapy
  Interventions: Device: Treatment plus Optimal Medical Therapy
- Optimal Medical Therapy (Active Comparator): Patients will be treated according to Optimal Medical Therapy
  Interventions: Other: Optimal Medical Therapy

INTERVENTIONS:
Device: Treatment plus Optimal Medical Therapy — Patients will be treated with the AeriSeal System in 2 subsegments in the upper lobes of each lung (4 subsegments total). 20mL of foam sealant will be injected via catheter into each subsegment selected for treatment. Patients will also receive Optimal Medical Therapy. Guidelines for prescribing medical treatment for emphysema have been published by the American Thoracic Society (ATS) and the National Heart Lung and Blood Institute/World Health Organization (NHLBI/WHO GOLD workshop summary).
  Other Names: AeriSeal System
  Arms: Treatment plus Optimal Medical Therapy
Other: Optimal Medical Therapy — Patients will receive Optimal Medical Therapy. Guidelines for prescribing medical treatment for emphysema have been published by the American Thoracic Society (ATS) and the National Heart Lung and Blood Institute/World Health Organization (NHLBI/WHO GOLD workshop summary).
  Arms: Optimal Medical Therapy

SUMMARY:
The purpose of this study is to demonstrate the safety and efficacy of AeriSeal System treatment plus optimal medical therapy compared in patients with advanced upper lobe predominant (ULP) heterogeneous emphysema.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent
2. Age ≥ 40 years
3. On optimal medical therapy* for more than 1 month
4. Advanced upper lobe predominant emphysema confirmed by CT scan
5. Two (2) subsegments appropriate for treatment in 2 different upper lobe segments in each lung based upon CT scan (total 4 available subsegments)
6. MRCD score of ≥ 2 post pulmonary rehab (using modified MRCD scale of 0-4)
7. 6MWT distance ≥ 150 m post pulmonary rehab
8. Spirometry 15 minutes after administration of a bronchodilator showing BOTH:

   1. FEV1 < 50% predicted
   2. FEV1/FVC ratio < 70%
9. Plethysmographic lung volumes showing BOTH:

   1. TLC > 100% predicted
   2. RV > 150% predicted
10. DLco ≥ 20% and ≤ 60% predicted
11. Blood gases and oxygen saturation showing BOTH:

    1. SpO2 ≥ 90% on ≤ 4 L/min supplemental O2
    2. PaCO2 < 65 torr
12. Smoking history of ≥ 20 pack-years with abstinence for 16 weeks

Exclusion Criteria:

1. Prior lung volume reduction surgery, lobectomy or pneumonectomy, or lung transplantation
2. Requirement for ventilator support (other than CPAP or BPAP for sleep apnea)
3. Three (3) or more COPD exacerbations requiring hospitalization within 1 year of Screening visit or a COPD exacerbation requiring hospitalization within 8 weeks
4. Use of systemic steroids > 20 mg/day or equivalent immunosuppressive agents, heparins, oral anticoagulants or investigational medications

   Exclusion Criteria (continued):
5. a-1 antitrypsin serum level of < 80 mg/dL (immunodiffusion) or < 11 µmol/L (nephelometry)
6. CT scan: Presence of any of the following radiologic abnormalities:

   1. Pulmonary nodule on CT scan greater than 1.0 cm in diameter
   2. Radiologic picture consistent with active pulmonary infection
   3. Significant interstitial lung disease
   4. Significant pleural disease
   5. Giant bullous disease
7. Clinically significant asthma
8. Clinically significant bronchiectasis
9. Pulmonary hypertension
10. Allergy or sensitivity to medications required to safely perform AeriSeal System treatment under general anesthesia or conscious (moderate procedural) sedation
11. Participation in an investigational study of a drug, biologic, or device not currently approved for marketing
12. Body mass index < 15 kg/m2 or > 35 kg/m2
13. Female patient pregnant or breast-feeding or planning to be pregnant in the next year
14. Any abnormal screening laboratory test result
15. Significant comorbidity including any of the following:

    1. HIV/AIDs
    2. Active malignancy
    3. Stroke or TIA within 12 months
    4. Myocardial infarction within 12 months
    5. Congestive heart failure within 12 months
16. Any condition that would interfere with the intent of the study or would make participation not in the best interest of the patient such as alcoholism, high risk for drug abuse or noncompliance in returning for follow-up visits

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | 12 Months
  Change from baseline measurement of FEV1

SECONDARY OUTCOMES:
Patient Reported Outcomes | 12 Months
  Change in Patient reported outcome from baseline.
Exercise Capacity | 12 months
  The change from baseline in Exercise Capacity
Radiological Changes | 12 months
  The radiological changes from baseline.

CONTACTS AND LOCATIONS:
Locations (40):
- United States (29):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Pulmonary Associates, Phoenix, Arizona
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Miami VA Healthcare System (accepting Miami VA patients only), Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - The University of Chicago Medicine, Chicago, Illinois
  - Presence Saint Joseph Medical Center, Joliet, Illinois
  - Illinois Lung Institute, Peoria, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veritas Clinical Specialties, Ltd., Topeka, Kansas
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Jamaica Hospital Medical Center, Jamaica, New York
  - South Nassau Communities Hospital, Oceanside, New York
  - Duke University Medical Center, Durham, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Kaiser Foundation Hospitals (accepting Kaiser patients only), Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of South Carolina School of Medicine, Columbia, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
- France (3):
  - CHU de Grenoble, Grenoble
  - CHU de Nice, Nice
  - Hôpital Maison Blanche, Reims
- University of Athens - Sotiria General Hospital, Athens, Greece
- Rabin Medical Center, Petah Tikva, Israel
- Azienda Ospedaliera Spedali Civili de Brescia, Brescia, Italy
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- Spain (4):
  - Hospital Universitari de Bellvitge, Barcelona
  - Fundación Jiménez Díaz, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario y Politécnico La Fe, Valencia

REFERENCES:
- [Derived] Come CE, Kramer MR, Dransfield MT, Abu-Hijleh M, Berkowitz D, Bezzi M, Bhatt SP, Boyd MB, Cases E, Chen AC, Cooper CB, Flandes J, Gildea T, Gotfried M, Hogarth DK, Kolandaivelu K, Leeds W, Liesching T, Marchetti N, Marquette C, Mularski RA, Pinto-Plata VM, Pritchett MA, Rafeq S, Rubio ER, Slebos DJ, Stratakos G, Sy A, Tsai LW, Wahidi M, Walsh J, Wells JM, Whitten PE, Yusen R, Zulueta JJ, Criner GJ, Washko GR. A randomised trial of lung sealant versus medical therapy for advanced emphysema. Eur Respir J. 2015 Sep;46(3):651-62. doi: 10.1183/09031936.00205614. Epub 2015 Apr 2. PMID 25837041